CLINICAL TRIAL: NCT01805284
Title: Pharmacokinetic and Pharmacodynamic Evaluation of Linezolid Administered Intravenously in MRSA-positive, Morbidly Obese Patients With Pneumonia
Acronym: UGENT_LIMOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012/788; 2012-005127-33 (EudraCT Number)
Record Dates: First submitted 2013-02-27; First posted 2013-03-06 (Estimated); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Pneumonia
Keywords: pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Linezolid (Experimental)
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Linezolid — 600 mg linezolid as a 1 hour controlled infusion (acceptable time frame is between 30 and 120 minutes), twice, at least 3 days.

SUMMARY:
The objectives of the study are:

(i) to evaluate the proportion of patients who attain a T>MIC (Minimum Inhibitory Concentration) of 100% and the time frame in which they do so. The investigators therefore plan to measure unbound linezolid trough concentrations before administration of the second, third, fourth and fifth dose. Furthermore, the investigators will assess the AUC0 - 24h/MIC in all study subjects. Therefore, multiple plasma samples will be drawn after the fourth or fifth dose, when steady state conditions are reached.

(ii) to describe the pharmacokinetic variability of unbound linezolid concentrations in this cohort using a population pharmacokinetic model and to assess the expected probability of target attainment (PTA) by MIC against MRSA.

Twenty adult, MRSA-positive, morbidly obese patients with clinically and radiologically documented pneumonia are to be included. Therefore, a multi-centre, international observational study is necessary. Given the specific target population this study is not feasible in a single-centre approach. The goal is to find up to 6 centres that anticipate including 3 to 4 patients in the study within a time frame of one year.

Included patients should receive at least 6 doses of linezolid. Linezolid must be administered intravenously (iv) over a one hour controlled infusion (with use of a volumetric infusion pump).

ELIGIBILITY:
* BMI >35
* Radiographically and clinically documented pneumonia and one of the following:

  * the patient is MRSA screen-positive and is as such at high risk for MRSA pneumonia (MIC for linezolid is known or possible to assess)
  * the patient has a baseline respiratory tract sample positive for MRSA; MRSA pneumonia is likely
  * empiric therapy without linezolid is initiated (no obvious indication for MRSA involvement), but the patient is switch to linezolid therapy once culture results demonstrate MRSA as pathogen. CAVE: the patients must be included in the study prior to the moment the first trough sample must be drawn. As such, patients becoming MRSA-positive after >1 dose of linezolid cannot be included in the study.
* Decision to start treatment with linezolid for at least 3 days (6 doses of 600 mg).
* Patient is colonized or infected with MRSA (at any site) and it must be possible to sent a fresh isolate to the central laboratory for microbiology.
* Written informed consent by the patient or his/her legal representative.

Exclusion:

Contraindications as described in the summary of product characteristics (SPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics/-dynamics of linezolid in blood samples: T>MIC of 100. | Over the course of 72 hours after the first administration of linezolid.
  A total of 17 blood samples will be collected over 72 hours after the first administration of linezolid, using a catheter.
  There will be evaluation of the proportion of patients who attain a T>MIC (Minimum Inhibitory Concentration) of 100% and the time frame in which they do so. The investigators therefore plan to measure unbound linezolid trough concentrations before administration of the second, third, fourth and fifth dose. Furthermore, the investigators will assess the AUC0 - 24h/MIC in all study subjects. Therefore, multiple plasma samples will be drawn after the fourth or fifth dose, when steady state conditions are reached
Pharmacokinetics/-dynamics of linezolid in urine samples. | During 12 hours after 6th or 7th administration of linezolid.
  This collection will be done using a catheter that was already in place, or will be collected in containers if no catheter is present at the time of this collection.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Vogelaers, Ph.D., M.D., Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium